CLINICAL TRIAL: NCT01695616
Title: A Phase III, Multicenter, Randomized, Double-blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Passiflora Incarnata and Isoflavona Combination in the Treatment of Climacteric Symptoms.
Brief Title: Efficacy and Safety of Passiflora Incarnata and Isoflavona Combination in the Treatment of Climacteric Symptoms
Acronym: Monalisa
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACH-SNT-03(01/12)
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Climacteric Syndrome
MeSH Terms: interventions — Bulk Drugs

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients enrolled in this arm will take a tablet twice a day
  Interventions: Drug: Placebo
- Passiflora incarnata and isoflavona combination (Active Comparator): Patients enrolled in this arm will take a tablet twice a day
  Interventions: Drug: Active drug

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: Active drug
  Arms: Passiflora incarnata and isoflavona combination

SUMMARY:
The purpose of this study is to evaluate the effects of Passiflora incarnata and Isoflavone combination in relieving the symptoms associated with Climacteric Syndrome.

DETAILED DESCRIPTION:
It is known that Hormone Therapy is recommended postmenopausal women to reduce menopausal symptoms and prevent osteoporosis frames and cardiovascular disease. However, only 30 to 40% of women still using hormone therapy.

One reason women do not continue or are reluctant to start Hormone Therapy is realizing that the prescription of hormones is not a natural situation. Therefore, there is an increased interest in the use and prescription of estrogen derived from plants, known as fitoestrogênios.

The development of a drug containing two standardized extracts was focused on two main symptoms of menopause: hot flashes and anxiety. This product comes from a longing for the doctors themselves can respond more promptly to patients who reach menopause and who already has a framework for mild to moderate anxiety.

Thus, to meet the woman who develops menopausal symptoms and that these two are highly prevalent during menopause, causing intense discomfort routine for this woman, was produced in association with Soy Passiflora aiming to control anxiety and hot flushes

ELIGIBILITY:
Inclusion Criteria:

* Female amenorrheic for at least one (1) year or surgical menopause since dosage of FSH ≥ 30 mIU / ml;
* Age greater than or equal to 40 and less than or equal to 65 years;
* Cytological examination colpo held at screening visit, Pap cytology classification with class I and II;
* By mammography BI-RADS classification (fourth edition) rated one (1) or two (2) performed at least six (6) months from the time of inclusion in the screening visit or if the research subject does not present a recent survey ;
* Line endometrial ≤ 8 mm by transvaginal ultrasound, performed at screening visit, in the case of subjects who have an intact uterus;

Exclusion Criteria:

* History of severe liver or renal disease at the discretion of the investigator;
* Hypertension stage III uncontrolled (SBP ≥ 180 mmHg or DBP ≥ 110 mmHg);
* Important cardiovascular disease such as coronary insufficiency or dilated cardiomyopathy advanced;
* Using estrogens, progestins, steroid or hormone replacement therapy (HRT) in the last 3 months;
* Estrogen-dependent neoplasia;
* Thromboembolic disorders for less than one year of screening visit;
* Anabolic drugs use or illicit drug use;
* Hemoglobin < 10 or > 17 g / dL;
* TSH < 0, 550 or > 4, 780 UUI / L;
* FT4 < 0.75 ηg / dL or > 1.8 ηg / dL;
* Patient that is chronically using MAO inhibitors (MAOIs) or levothyroxine

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Menopause Rating Scale - MRS | 104 days

SECONDARY OUTCOMES:
Kuppperman-Blatt index | 90 days
MRS scale | 90 days
MENQOL | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- ISBEM, São Paulo, São Paulo, Brazil